CLINICAL TRIAL: NCT04690933
Title: Real-life Observatory of Efficacy and Resistance to Anti CMV Molecules in Stem Cell Recipients
Brief Title: AntiCMV molécules Monitoring in Real-life in Stem Cell Recipients
Acronym: NAViRe
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18_0011 (NAViRe)
Record Dates: First submitted 2020-09-14; First posted 2020-12-31 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2020-09

CONDITIONS: Hematopoietic Stem Cell Transplantation; Cytomegalovirus Infections; Antivirals; Antiviral Drug Resistance
Keywords: Hematopoietic Stem Cell Transplantation; Cytomegalovirus Infections; Antivirals; Antiviral Drug Resistance
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples related to the cohort :
  One blood sample from the donor (only familial donors) for genetic SNPs analysis.
  5 samples: D-8 (conditioning), D20, D100 (+/- 10 days), D200 (+/- 10 days), 1 year : 1 tube of 7ml of whole blood on EDTA: Biobanking of whole blood for genetic SNPs analysis (D-8) of specific transporters for GCV, and of plasma for TTV viral load at all times. Conservation of viral load monitoring remnants at the center's virology laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multicentric NAViRe cohort with biocollection: The National Reference Center (CNR) for cytomegalovirus with the French Society for Medullary Transplantation and Cell Therapy (SFGM-TC) has set up a surveillance cohort of allografted patients (NAViRe cohort) receiving, as prevention or treatment, Anti-Cytomegalovirus (Anti-CMV) molecules, "new or less recent", thus allowing the development of a new observatory evaluating in real life the potentials of these drugs in terms of efficacy, emergence of resistance, tolerance and morbidity and mortality associated with CMV infection.This work is useful to propose recommendations on management strategies, in particular for the most at-risk patients i.e. CMV-seropositive recipients and allows the emergence of an real-life observatory of efficacy and resistance to anti CMV molecules in stem cell recipients.
  Interventions: Other: Real-life observatory of efficacy and resistance to anti CMV molecules in stem cell recipients

INTERVENTIONS:
Other: Real-life observatory of efficacy and resistance to anti CMV molecules in stem cell recipients — Signing of consent at the time of the pre-transplant consultation (1 month before grafting). Inclusion of patients during conditioning (around D-8 of transplantation). Samples related to the cohort:one blood sample from the donor (only familial donors) for genetic SNPs analysis. 5 samples: D-8, D20, D100, D200 (+/-10 days), 1 year : 1 tube of 7ml of whole blood on EDTA: Biobanking of whole blood for genetic SNPs analysis (D-8) of specific transporters for GCV, and of plasma for TTV viral load at all times. In routine care:samples taken in the event of a therapeutic escape (2 x 7 ml EDTA tubes, for resistance genotype, and ganciclovir dosage, 3 x 1 ml for Quantiferon CMV, according to CNR Herpesvirus recommendations. 1 x Paxgene tube (2.5 ml) for subsequent CMV genomic and transcriptomic studies. Cell preservation plasma and whole blood for biocollection (2 tubes EDTA de 7ml). Samples stored by the centers' virology laboratories are periodically sent to the CNR for analysis.

SUMMARY:
Cytomegalovirus (CMV) is a ubiquitous herpesvirus that represent a major cause of morbidity in haematopoietic stem cell transplants (HSCT) recipients, mostly through reactivation of the recipient's virus.

If left untreated, 40 to 80% of patients will develop CMV infection, leading to CMV disease in 30 to 35 % patients, and associated with considerable morbi-mortality. Interstitial pneumonia is the most severe and specific manifestation, although CMV replication by itself has also indirect effects such as triggering graft versus host disease and increasing immunosuppression. The current burden of CMV infection increases by 25 to 30% the cost of the graft in France. This also includes the burden for refractory - infections, that represent up to 13% of recipients with CMV infection, including 3% of cases with virological resistance in France (data from the Reference Center cohorts).

Ganciclovir, or valganciclovir preemptive treatment, guided by CMV viral load follow-up allowed significant reduction of CMV disease to 2-6% but did not prevent CMV indirect effects. In addition, hematotoxicity can compromise post-transplant haematological reconstitution, thus preventing its use as prophylaxis in France. Foscarnet, iv-administered and nephrotoxic, remains less used. There is thus a high expectation from less toxic molecules for prophylaxis The development letermovir recently available for prophylaxis of CMV infection in high risk patients will modify the patients care and follow-up. This new molecule targeting CMV terminases (developed by Merck) was recently marketed in France (Jan 2020). However, the analysis of the letermovir phase III study and further publications show that the risk of emergence of resistance is low, but may occur in case of breakthrough and thus post AMM monitoring is required.

A "real-life" evaluation of these new molecules in terms of efficacy, emergence of resistance, tolerance and morbimortality related to CMV infection, is useful, to propose recommendations on management strategies, in particular for the most at-risk patients i.e. CMV-seropositive recipients. To this purpose, the National Reference Center in collaboration with the French Society for marrow graft and cell therapy (SFGMTC) set up a cohort of surveillance of allografted patients, receiving, in prevention or treatment, old and new molecules.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is a ubiquitous herpesvirus that represent a major cause of morbidity in haematopoietic stem cell transplants (HSCT) recipients, mostly through reactivation of the recipient's virus.

If left untreated, 40 to 80% of patients will develop CMV infection, leading to CMV disease in 30 to 35 % patients, and associated with considerable morbi-mortality. Interstitial pneumonia is the most severe and specific manifestation, although CMV replication by itself has also indirect effects such as triggering graft versus host disease and increasing immunosuppression. The current burden of CMV infection increases by 25 to 30% the cost of the graft in France. This also includes the burden for refractory - infections, that represent up to 13% of recipients with CMV infection, including 3% of cases with virological resistance in France (data from the Reference Center cohorts).

Ganciclovir, or valganciclovir preemptive treatment, guided by CMV viral load follow-up allowed significant reduction of CMV disease to 2-6% but did not prevent CMV indirect effects. In addition, hematotoxicity can compromise post-transplant haematological reconstitution, thus preventing its use as prophylaxis in France. Foscarnet, iv-administered and nephrotoxic, remains less used. There is thus a high expectation from less toxic molecules for prophylaxis The development letermovir recently available for prophylaxis of CMV infection in high risk patients will modify the patients care and follow-up. This new molecule targeting CMV terminases (developed by Merck) was recently marketed in France (Jan 2020). However, the analysis of the letermovir phase III study and further publications show that the risk of emergence of resistance is low, but may occur in case of breakthrough and thus post AMM monitoring is required.

A "real-life" evaluation of these new molecules in terms of efficacy, emergence of resistance, tolerance and morbimortality related to CMV infection, is useful, to propose recommendations on management strategies, in particular for the most at-risk patients i.e. CMV-seropositive recipients. To this purpose, the National Reference Center in collaboration with the French Society for marrow graft and cell therapy (SFGMTC) set up a cohort of surveillance of allografted patients, receiving, in prevention or treatment, old and new molecules.

ELIGIBILITY:
Inclusion Criteria :

• Candidate (adult) for an allograft of hematopoietic stem cells for which a decision of transplant is made and willing to participate in the cohort.

Exclusion Criteria :

* CMV-seronegative patient receiving a negative CMV donor graft ;
* Patient having signed the consent but not grafted ;
* Patient included in a clinical study on an anti-CMV molecule ;
* Non-insured social patient ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidate (adult) for an allograft of hematopoietic stem cells for which a decision of transplant is made and willing to participate in the cohort.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
CMV infection according to criteria defined by the European EBMT group (Ljungman et al., 2017). | between Day-30 and Day -8
  CMV detection (CMV DNAemia or antigen detection) in any body fluid or tissue specimen
CMV infection according to criteria defined by the European EBMT group (Ljungman et al., 2017). | between Day-8 and Day 0
  CMV detection (CMV DNAemia or antigen detection) in any body fluid or tissue specimen
CMV infection according to criteria defined by the European EBMT group (Ljungman et al., 2017). | at Day20
  CMV detection (CMV DNAemia or antigen detection) in any body fluid or tissue specimen
CMV infection according to criteria defined by the European EBMT group (Ljungman et al., 2017). | at Day100
  CMV detection (CMV DNAemia or antigen detection) in any body fluid or tissue specimen
CMV infection according to criteria defined by the European EBMT group (Ljungman et al., 2017). | at Day 200 (Month 6)
  CMV detection (CMV DNAemia or antigen detection) in any body fluid or tissue specimen
CMV infection according to criteria defined by the European EBMT group (Ljungman et al., 2017). | Month12
  CMV detection (CMV DNAemia or antigen detection) in any body fluid or tissue specimen
CMV infection according to criteria defined by the European EBMT group (Ljungman et al., 2017). | Month24
  CMV detection (CMV DNAemia or antigen detection) in any body fluid or tissue specimen

SECONDARY OUTCOMES:
Uses of anti-CMV molecules : preemptive treatment | at Day200
  % of patients having received preemptive treatment
Uses of anti-CMV molecules : prophylaxis | at Day200
  % of patients having received prophylaxis
Uses of anti-CMV molecules : curative treatment | at Day200
  % of patients having received curative treatment
Uses of anti-CMV molecules | at Day200
  Cumulative duration of exposure (number of day) for each drug administered
Uses of anti-CMV molecules : preemptive treatment | at Month12
  % of patients having received preemptive treatment
Uses of anti-CMV molecules : prophylaxis | at Month12
  % of patients having received prophylaxis
Uses of anti-CMV molecules : curative treatment | at Month12
  % of patients having received curative treatment
Uses of anti-CMV molecules | at Month12
  Cumulative duration of exposure (number of day) for each drug administered
Uses of anti-CMV molecules : preemptive treatment | at Month24
  % of patients having received preemptive treatment
Uses of anti-CMV molecules : prophylaxis | at Month24
  % of patients having received prophylaxis
Uses of anti-CMV molecules : curative treatment | at Month24
  % of patients having received curative treatment
Uses of anti-CMV molecules | at Month24
  Cumulative duration of exposure (number of day) for each drug administered
Incidence of the non-response and resistance to antivirals with risk factors associated (virological, pharmacological, immunological). Criteria recently published by Chemaly et al. CID 2018 will be used to classify cases in | at Month12
  Criteria recently published by Chemaly et al. CID 2018 will be used to classify cases in :
  * Refractory CMV infection CMV viremia that increases after at least 2 wk of appropriately dosed antiviral therapy.
  * Probable refractory CMV infection : persistent viral load after at least 2 wk of appropriately dosed antiviral therapy.
  * Refractory CMV end organ disease : worsening in signs and symptoms or progression into end-organ disease after at least 2 wk of appropriately dosed antiviral therapy.
  * Probable refractory CMV end-organ disease : lack of improvement in signs and symptoms after at least 2 wk of appropriately dosed antiviral drugs.
  * Antiviral drug resistance : viral genetic alteration that decreases susceptibility to one or more antiviral drugs.
  Resistance : presence of a resistance-related mutation by resistance genotyping of UL97, UL54, UL56, UL89, UL27 genes, carried out or validated by the Limoges Herpesviruses reference laboratory. In blood or any other sample.
Incidence of the non-response and resistance to antivirals with risk factors associated (virological, pharmacological, immunological). Criteria recently published by Chemaly et al. CID 2018 will be used to classify cases in | at Month24
  Criteria recently published by Chemaly et al. CID 2018 will be used to classify cases in :
  * Refractory CMV infection CMV viremia that increases after at least 2 wk of appropriately dosed antiviral therapy.
  * Probable refractory CMV infection : persistent viral load after at least 2 wk of appropriately dosed antiviral therapy.
  * Refractory CMV end organ disease : worsening in signs and symptoms or progression into end-organ disease after at least 2 wk of appropriately dosed antiviral therapy.
  * Probable refractory CMV end-organ disease : lack of improvement in signs and symptoms after at least 2 wk of appropriately dosed antiviral drugs.
  * Antiviral drug resistance : viral genetic alteration that decreases susceptibility to one or more antiviral drugs.
  Resistance : presence of a resistance-related mutation by resistance genotyping of UL97, UL54, UL56, UL89, UL27 genes, carried out or validated by the Limoges Herpesviruses reference laboratory. In blood or any other sample.
Adverse effects leading to interruption of treatment | at Month12
  Incidence of treatment emergent adverse event as assessed by interruption of treatment
Adverse effects leading to interruption of treatment | at Month24
  Incidence of treatment emergent adverse event as assessed by interruption of treatment
CMV related mortality | at Month12
  Number of patients who died from CMV related desease
CMV related mortality | at Month24
  Number of patients who died from CMV related desease
CMV associated morbidity : delay engraftment | at Month12
  number of days bettwen graft and engraftment
CMV associated morbidity : GVHD | at Month12
  Incidence of GVHD
CMV associated morbidity : CMV infection/disease | at Month12
  Incidence of CMV infection/disease (infection or disease will be combined to report this outcome).
  CMV infection : positive diagnostic test (CMV culture, antigen detection or CMV PCR), in any body fluid or tissue, in the absence of symptoms.
  CMV disease : CMV infection associated with end-organ disease (clinical signs and oriented virological diagnosis).
CMV associated morbidity : delay engraftment | at Month24
  number of days bettwen graft and engraftment
CMV associated morbidity : GVHD | at Month24
  Incidence of GVHD
CMV associated morbidity : CMV infection/disease | at Month24
  Incidence of CMV infection/disease (infection or disease will be combined to report this outcome).
  CMV infection : positive diagnostic test (CMV culture, antigen detection or CMV PCR), in any body fluid or tissue, in the absence of symptoms.
  CMV disease : CMV infection associated with end-organ disease (clinical signs and oriented virological diagnosis).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal TURLURE, Principal Investigator — Service d'Hématologie Clinique et de Thérapie Cellulaire
Locations (16):
- France (16):
  - CHU de LIMOGES, Limoges, Limoges
  - CHU, Amiens
  - CHU, Angers
  - CHU, Besançon
  - CHU, Bordeaux
  - CHU, Caen
  - CHU, Clermont-Ferrand
  - CHU, Grenoble
  - HCL, Lyon
  - CHU, Montpellier
  - CHU, Nancy
  - APHP, Paris
  - CHU, Poitiers
  - CHU, Rouen
  - CHU, Saint-Etienne
  - CHU, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ljungman P, Boeckh M, Hirsch HH, Josephson F, Lundgren J, Nichols G, Pikis A, Razonable RR, Miller V, Griffiths PD; Disease Definitions Working Group of the Cytomegalovirus Drug Development Forum. Definitions of Cytomegalovirus Infection and Disease in Transplant Patients for Use in Clinical Trials. Clin Infect Dis. 2017 Jan 1;64(1):87-91. doi: 10.1093/cid/ciw668. Epub 2016 Sep 28. PMID 27682069
- [Background] Chemaly RF, Chou S, Einsele H, Griffiths P, Avery R, Razonable RR, Mullane KM, Kotton C, Lundgren J, Komatsu TE, Lischka P, Josephson F, Douglas CM, Umeh O, Miller V, Ljungman P; Resistant Definitions Working Group of the Cytomegalovirus Drug Development Forum. Definitions of Resistant and Refractory Cytomegalovirus Infection and Disease in Transplant Recipients for Use in Clinical Trials. Clin Infect Dis. 2019 Apr 8;68(8):1420-1426. doi: 10.1093/cid/ciy696. PMID 30137245
- [Background] Billat PA, Ossman T, Saint-Marcoux F, Essig M, Rerolle JP, Kamar N, Rostaing L, Kaminski H, Fabre G, Otyepka M, Woillard JB, Marquet P, Trouillas P, Picard N. Multidrug resistance-associated protein 4 (MRP4) controls ganciclovir intracellular accumulation and contributes to ganciclovir-induced neutropenia in renal transplant patients. Pharmacol Res. 2016 Sep;111:501-508. doi: 10.1016/j.phrs.2016.07.012. Epub 2016 Jul 9. PMID 27402191
- [Background] Marty FM, Ljungman P, Chemaly RF, Maertens J, Dadwal SS, Duarte RF, Haider S, Ullmann AJ, Katayama Y, Brown J, Mullane KM, Boeckh M, Blumberg EA, Einsele H, Snydman DR, Kanda Y, DiNubile MJ, Teal VL, Wan H, Murata Y, Kartsonis NA, Leavitt RY, Badshah C. Letermovir Prophylaxis for Cytomegalovirus in Hematopoietic-Cell Transplantation. N Engl J Med. 2017 Dec 21;377(25):2433-2444. doi: 10.1056/NEJMoa1706640. Epub 2017 Dec 6. PMID 29211658
- [Background] Robin C, Hemery F, Dindorf C, Thillard J, Cabanne L, Redjoul R, Beckerich F, Rodriguez C, Pautas C, Toma A, Maury S, Durand-Zaleski I, Cordonnier C. Economic burden of preemptive treatment of CMV infection after allogeneic stem cell transplantation: a retrospective study of 208 consecutive patients. BMC Infect Dis. 2017 Dec 5;17(1):747. doi: 10.1186/s12879-017-2854-2. PMID 29207952
- [Result] Billat PA, Woillard JB, Essig M, Sauvage FL, Picard N, Alain S, Neely M, Marquet P, Saint-Marcoux F. Plasma and intracellular exposure to ganciclovir in adult renal transplant recipients: is there an association with haematological toxicity? J Antimicrob Chemother. 2016 Feb;71(2):484-9. doi: 10.1093/jac/dkv342. Epub 2015 Nov 3. PMID 26538506
- [Result] Kotton CN, Kumar D, Caliendo AM, Huprikar S, Chou S, Danziger-Isakov L, Humar A; The Transplantation Society International CMV Consensus Group. The Third International Consensus Guidelines on the Management of Cytomegalovirus in Solid-organ Transplantation. Transplantation. 2018 Jun;102(6):900-931. doi: 10.1097/TP.0000000000002191. PMID 29596116